CLINICAL TRIAL: NCT00001922
Title: Sensory Function in Idiopathic Voice Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990009; 99-N-0009
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-09-14

CONDITIONS: Phonation Disorder; Spastic Dysphonia; Voice Disorder
Keywords: Evoked Response; Spasmodic Dysphonia; Aerodynamic; Vibration; Laryngeal; Voice Disorders; Laryngeal Brainstem Evoked Responses; Long-latency Responses; Muscular Tension Dysphonia
MeSH Terms: conditions — Dysphonia; Voice Disorders; Laryngeal Diseases

SUMMARY:
This research study is designed to improve understanding about voice disorders that are due to uncontrolled muscle contractions affecting the voice box. The type of voice disorder depends on which muscles of the voice box are involved. Abductor spasmodic dysphonia may lead to a weak voice. Adductor spasmodic dysphonia may result in a strangled voice. Muscular tension dysphonia may lead to a strained voice. Some of the major goals of the study are to;

1. understand how sensation from the voice box affects voice and speech production
2. develop better ways to diagnose sensation abnormalities affecting the voice box
3. determine if patients with voice disorders differ from persons without voice disorders in the way they respond to sensory information from their voice box

Researchers believe that by understanding better how sensations of the voice box are presented and how the muscles in the larynx respond to those sensations they will be able to develop better treatments for patients suffering from voice disorders. ...

DETAILED DESCRIPTION:
Study Aim One: To develop and validate objective procedures for quantifying efferent responses to non-invasive laryngeal mechanical and aerodynamic stimulation.

Study Aim Two: To develop and validate an objective test of brain stem evoked responses to laryngeal stimulation using electrical stimulation of the superior laryngeal nerve.

Study Aim Three: To determine whether individuals with idiopathic voice disorders have abnormal conditioning of their responses to laryngeal mechanical and aerodynamic stimulation.

Study Aim Four: To determine whether individuals with idiopathic voice disorders have abnormal brain stem responses to laryngeal stimuli.

Study Aim Five: To evaluate whether sensory input plays a role in symptom generation in laryngeal motor control disorders, temporary bilateral ISLN blockade will be used in idiopathic voice disorders.

Study Aim Six: To evaluate whether the central pathophysiology involved in motor responses to sensory stimulation are altered by botulinum toxin injection in individuals with spasmodic dysphonia.

Study Aim Seven: To evaluate central responses to laryngeal afferent stimulation in normal volunteers and patients with idiopathic voice disorders at rest and during vocalization using magnetoencephalography.

These studies will develop improved non-invasive techniques for the diagnosis of laryngeal sensory disorders and will determine if abnormalities in sensory feedback modulation are involved in idiopathic voice disorders. Such findings will lead to improved understanding of the pathophysiology and differential diagnosis of idiopathic voice disorders and may ultimately improve treatment approaches to these disorders.

ELIGIBILITY:
* INCLUSION CRITERIA - Normal Volunteers:
* Normal volunteers between the ages of 20 and 80 years of age will be selected after a screening examination.
* Subjects will be without cardiac, pulmonary, neurological, otolaryngological, psychiatric or speech and hearing problems as determined by medical history and examination by an otolaryngologist.
* None of the subjects included for study will have a reduction in the range of vocal fold movement during non-speech tasks such as whistling suggesting either paralysis or paresis, joint abnormality or neoplasm.

EXCLUSION CRITERIA - Normal Volunteers:

* Any patient with a history of airway obstruction will be excluded from the study.
* No smokers or tobacco users will be included in the study.
* Subjects with a history of a psychiatric disorder, under the care of a psychiatrist, or on medications for treatment of a psychiatric disorder will be excluded from study. Examples of psychiatric disorders to be excluded are: somatoform disorders, conversion disorders, currently under treatment for a major depression, or a history of schizophrenia or a bipolar disorder. However, a history of a previous episode of a minor reactive depression would not exclude a person from participation.

Any individual with: 1) an implant or surgical clip - implanted neural stimulator, implanted cardiac pacemaker or autodefibrillator, cochlear implant, ocular implant, aneurysm clip, artificial heart valve, insulin pump, orthopedic pins or prosthesis: 2) a foreign body - metal shavings, shrapnel, orthodontic braces, tattoos or permanent eye liner; and/or, 3) any other implanted device or foreign body not listed above that is possibly ferromagnetic will also be excluded from study seven because of contraindications for magnetic resonance imaging.

INCLUSION CRITERIA - Patients with Spasmodic Dysphonia:

* Symptoms present during speech and not apparent at rest.
* Symptoms less evident during whisper, singing or falsetto.
* Symptoms become worse with prolonged speaking, practice or anxiety.
* Reflexive and emotional aspects of voice function are unaffected, such as coughing, laughter or crying.

EXCLUSION CRITERIA - Patients with Spasmodic Dysphonia:

* Any patient with a history of airway obstruction will be excluded from the study. Structural abnormalities affecting the larynx such as vocal fold nodules, polyps, carcinoma, cysts, contact ulcers, or inflammation (laryngitis).
* Reduction in vocal fold movement range during non-speech tasks such as whistling which would suggest either paralysis or paresis, joint abnormality or neoplasm.
* No smokers or tobacco users will be included in the study.
* Subjects with a history of a psychiatric disorder, under the care of a psychiatrist, or on medications for treatment of a psychiatric disorder will be excluded from study. Examples of psychiatric disorders to be excluded are: somatoform disorders, conversion disorders, currently under treatment for a major depression, or a history of schizophrenia or a bipolar disorder. However, a history of a previous episode of a minor reactive depression would not exclude a person from participation.
* Although patients with neurological disorders are excluded, certain focal dystonias which occasionally occur simultaneously with spasmodic dysphonia, will not automatically exclude a patient from participating. The determination will be made at the discretion of the Laryngeal and Speech Section Team.
* Although structural abnormalities of the larynx will cause a patient to be excluded, those that have had previous laryngeal surgery will not automatically be disqualified if they remain measurably symptomatic with their voice disorder. The determination will be made at the discretion of the Laryngeal and Speech Section Team.
* Patients whose symptoms vary during their initial interview, and/or who report periods of symptom remission and are atypical of spasmodic dysphonia will not be included.
* Patients with whispering aphonia or complete aphonia will not be included.
* Patients with a constant voice quality abnormality will not be included.
* Patients with muscular tension dysphonia will be included in a separate subject group and not included in spasmodic dysphonia.
* Spasmodic dysphonia and muscular tension dysphonia are disorders of adult onset usually first occurring after 40 years of age, therefore, we do not plan to include children in this study.

INCLUSION CRITERIA - Patients with Adductor SD:

* Intermittent strained hoarseness and uncontrolled voice breaks or changes in pitch during vowels in speech.
* Symptoms most easily heard on vowels, liquids (r and l) or semivowel sounds (w and y).
* Intermittent hyperadduction of the vocal folds interfering with air flow through the folds during vowels in speech, stopping vocal fold vibration, and resulting in voice interruptions or breaks. When the hyperadduction is less severe, voicing may become strained or a rapid change in pitch may occur. In the milder forms of the disorder, only intermittent irregular catches will be heard in the voice on a vowel every couple of sentences. In the moderate form, the voice is constantly breaking or bursting as the patient tries to force air through excessively tight vocal folds. The speech has intermittent hoarseness as well. In the most severe form, individuals have a constant strained hoarseness and reduced volume because very little air can be forced through the vocal folds. In such individuals voice may be heard only at the end of sentences as the vocal folds release at the end of speech phrases. The speech is excessively slow, tight and effortful.

INCLUSION CRITERIA - Patients with Abductor SD:

* Prolonged vocal fold opening during voiceless consonants with excessive breathiness as individuals experience difficulties in closing the vocal folds to produce vowels following voiceless consonants (p, t, k, s, f, h, th). Sounds such as (s, h or k) when coming just before open vowels such as (ah and uh) as in home, coffee and puppy are usually most affected.
* A breathy voice quality, uncontrolled pitch elevations on vowel initiation, difficulty coordinating breathing with speech, and complaints of excessive air loss while speaking. These individuals usually have similar problems in singing but normal laughter and coughing. In the milder forms only intermittent prolongations of a few voiceless consonants are heard. In the more severe forms more voiceless consonants are affected, speech initiation becomes more difficult and voice becomes breathy. In the most severe forms of both adductor and abductor spasmodic dysphonia, individuals may resort to whispering which is less affected and much less effortful.

EXCLUSION CRITERIA - Patients with Adductor SD:

* Any patient with a history of airway obstruction will be excluded from the study.
* No smokers or tobacco users will be included in the study.
* Patients with cardiac, pulmonary, neurological, otolaryngological, psychiatric or speech and hearing problems as determined by medical history and examination by an otolaryngologist.
* Structural abnormalities affecting the larynx such as vocal fold nodules, polyps, carcinoma, cysts, contact ulcers, or inflammation (laryngitis).
* Reduction in vocal fold movement range during non-speech tasks such as whistling which would suggest either paralysis or paresis, joint abnormality or neoplasm.
* Patients whose symptoms vary during their initial interview, and/or who report periods of symptom remission and are atypical of spasmodic dysphonia will not be included.
* Patients with whispering aphonia or complete aphonia will not be included.
* Patients with muscular tension dysphonia will be included in a separate subject group and not included in spasmodic dysphonia.

EXCLUSION CRITERIA - Patients with Abductor SD:

* Any patient with a history of airway obstruction will be excluded from the study.
* No smokers or tobacco users will be included in the study.
* Patients with cardiac, pulmonary, neurological, otolaryngological, psychiatric or speech and hearing problems as determined by medical history and examination by an otolaryngologist.
* Structural abnormalities affecting the larynx such as vocal fold nodules, polyps, carcinoma, cysts, contact ulcers, or inflammation (laryngitis).
* Reduction in vocal fold movement range during non-speech tasks such as whistling which would suggest either paralysis or paresis, joint abnormality or neoplasm.
* Patients whose symptoms vary during their initial interview, and/or who report periods of symptom remission and are atypical of spasmodic dysphonia will not be included.
* Patients with whispering aphonia or complete aphonia will not be included.
* Patients with muscular tension dysphonia will be included in a separate subject group and not included in spasmodic dysphonia.

INCLUSION CRITERIA - Patients with Muscular Tension Dysphonia:

1. Increased phonatory muscle tension in the paralaryngeal and suprahyoid muscles on palpation.
2. Constant elevation of the larynx in the neck during speech.
3. A consistent hypertonic laryngeal posture for phonation, either an open posterior glottic chink between the arytenoid cartilages on phonation, an anterior-posterior squeeze (pinhole posture) or ventricular hyperadduction.
4. A normal appearing larynx.

EXCLUSION CRITERIA - Patients with Muscular Tension Dysphonia:

1. Cardiac, pulmonary, neurological, otolaryngological, psychiatric or speech and hearing problems as determined by medical history and examination by a physician. Any patient with a history of airway obstruction will be excluded from the study.
2. Reduction in the range of vocal fold movement during non-speech tasks such as whistling suggesting either paralysis or paresis, joint abnormality or neoplasm.
3. Intermittent symptoms during their initial interview, reports of periods of symptom remission or spasmodic breaks in voicing typical or either adductor or abductor spasmodic dysphonia.
4. A 30 dB HL screening between 500 and 3000 Hz will be conducted if subjects report difficulty following spoken instructions and a history of hearing loss or significant noise exposure.
5. No smokers or tobacco users will be included in the study.
6. Exclude mucosal changes such as vocal nodules or polyps.
7. Subjects with a history of a psychiatric disorder, under the care of a psychiatrist, or on medications for treatment of a psychiatric disorder will be excluded from study. Examples of psychiatric disorders to be excluded are: somatoform disorders, conversion disorders, currently under treatment for a major depression, or a history of schizophrenia or a bipolar disorder. However, a history of a previous episode of a minor reactive depression would not exclude a person from participation.

OTHER EXCLUSION CRITERIA:

Subjects will be excluded if they have a history of rheumatic fever, mitral valve prolapse or cardiac arrhythmias, as determined by medical history, physical and EKG.

Individuals who might be at risk for endocarditis will be excluded.

All patients over the age of 40 years of age will have an electrocardiogram on the day of the study and if there are any abnormalities they will not be allowed to participate.

Pregnancy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370
Dates: Start 1998-11-05; Primary Completion 2009-09-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sant'Ambrogio G, Mathew OP. Laryngeal receptors and their reflex responses. Clin Chest Med. 1986 Jun;7(2):211-22. PMID 3522068
- [Background] Sant'Ambrogio G, Anderson JW, Sant'Ambrogio FB, Mathew OP. Response of laryngeal receptors to water solutions of different osmolality and ionic composition. Respir Med. 1991 Jan;85 Suppl A:57-60. doi: 10.1016/s0954-6111(06)80256-8. PMID 2034837
- [Background] Hansson L, Wollmer P, Dahlback M, Karlsson JA. Regional sensitivity of human airways to capsaicin-induced cough. Am Rev Respir Dis. 1992 May;145(5):1191-5. doi: 10.1164/ajrccm/145.5.1191. PMID 1586064